CLINICAL TRIAL: NCT06103422
Title: Evaluation of Change in Taste Sense After Orthognathic Surgery
Brief Title: Change in Taste Sensation After Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yağmur Malkoc (Other)
Collaborators: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor-Investigator, Yağmur Malkoc, DDS (Doctor of Dental Surgery), Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IstanbulMUH-DF-YM-01
Record Dates: First submitted 2023-10-23; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Orthognathic Surgery; Altered Taste
Keywords: Gustation; Taste sense
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Streaming of patients and administration of tests (Experimental): 35 patients who met the inclusion criteria were divided into surgical groups. Patients with indications for upper jaw surgery were divided into Le Fort I operation, patients with lower jaw surgery were divided into Sagittal Split Ramus operation, and double jaw surgery groups. Localized taste tests and whole-mouth taste tests were applied to the patients.
  Interventions: Diagnostic Test: Whole mouth taste tests; Diagnostic Test: Localized taste tests
- Repetition of tests at certain intervals (Experimental): Gustatory functions were evaluated by administering localized taste tests and whole mouth taste tests preoperatively and at postoperative 1st, 3rd, and 6th months.
  Interventions: Diagnostic Test: Whole mouth taste tests; Diagnostic Test: Localized taste tests

INTERVENTIONS:
Diagnostic Test: Whole mouth taste tests — Patients who underwent Le Fort I osteotomy, Sagittal Split Ramus Osteotomy, and Bimaxillary Surgeries were asked to identify the quality of 4 basic taste modalities preoperatively and at postoperative 1st, 3rd, and 6th months by administering whole mouth taste tests. In the whole mouth taste test, one ml of the specific solution was drawn into the syringe and sprayed into the mouth of the patient circularly. After each administration, patients spat out the solutions and reported whether they perceived any taste and, if so, which taste it was.
Diagnostic Test: Localized taste tests — Patients who underwent Le Fort I osteotomy, Sagittal Split Ramus Osteotomy, and Bimaxillary Surgeries were asked to identify the quality of 4 basic taste modalities preoperatively and at postoperative 1st, 3rd, and 6th months by administering localized taste tests. In the localized mouth taste test, the highest concentration solution of one of the four flavors was administered. In each application, 0.25 ml of solution was absorbed on a sterile cotton swab and applied on 6 test areas on the palate and tongue.
  Other Names: Spatial taste test

SUMMARY:
Orthognathic surgery refers to jaw operations that can be performed on the upper jaws (Le Fort I osteotomy) and lower jaws (Sagittal Split Ramus osteotomy). In orthognathic surgery practice, taste perception could be affected by potential damage to peripheral nerves that conduct chemosensory information regarding gustation from the palate and tongue. This study aimed to evaluate the changes in the sense of taste after Le Fort I osteotomy, Sagittal Split Ramus osteotomy, and bimaxillary surgery.

DETAILED DESCRIPTION:
The subjects were orthognathic surgery patients with facial skeletal deformities who applied to the Department of Oral and Maxillofacial Surgery. Thirty-five patients, aged 17-42 years, gustatory functions were evaluated by administering localized taste tests and whole mouth taste tests preoperatively and at postoperative 1st, 3rd, and 6th months. In the tests, solutions containing sucrose for a sweet taste, sodium chloride for a salty taste, citric acid for a sour taste, and quinine hydrochloride for a bitter taste were used. Patients were compared between the operation group they were in and between operation groups.

ELIGIBILITY:
Inclusion Criteria:

* dentofacial deformity
* American Society of Anesthesiologists category 1 or 2

Exclusion Criteria:

* zinc, iron, and/or vitamin deficiencies
* oncological, neurological, endocrinological, and rheumatological diseases
* chronic drug use due to systemic disease
* smokers
* history of chemotherapy and radiotherapy to the head and neck region, orthognathic surgery, maxillofacial trauma, and damage to the nerves related to the taste sensation

Ages: 17 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Taste recognition threshold | Six months
  The solutions were administered in increasing concentrations, starting from the lowest concentration up to the highest concentration until the patient perceived any taste. The lowest concentration at which the patient correctly perceived the administered taste was defined as the "taste recognition threshold. Taste recognition threshold is the primer outcome for whole-mouth taste tests.
Taste intensity rating | Six months
  The patients were instructed to focus on the perceived taste without closing their mouths and asked to identify the taste and rate the intensity of the taste using a scale ranging between 0 'no taste' and 9 'strongest taste', after each administration. Taste intensity rating is the primer outcome for localized taste tests.

CONTACTS AND LOCATIONS:
Overall Officials: Sina UÇKAN, Study Director — Medipol University
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medipol University, Istanbul, Bağcılar, Istanbul
  - Istanbul Medipol University, Istanbul, Fatih

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowe DC, Gruber EA, McLeod NM. Nerve injury associated with orthognathic surgery. Part 1: UK practice and motor nerve injuries. Br J Oral Maxillofac Surg. 2016 May;54(4):362-5. doi: 10.1016/j.bjoms.2016.01.026. Epub 2016 Feb 28. PMID 26935213
- [Background] Gent JF, Shafer DM, Frank ME. The effect of orthognathic surgery on taste function on the palate and tongue. J Oral Maxillofac Surg. 2003 Jul;61(7):766-73. doi: 10.1016/s0278-2391(03)00152-6. PMID 12856248
- [Background] Al-Din OF, Coghlan KM, Magennis P. Sensory nerve disturbance following Le Fort I osteotomy. Int J Oral Maxillofac Surg. 1996 Feb;25(1):13-9. doi: 10.1016/s0901-5027(96)80005-1. PMID 8833294
- [Background] Ylikontiola L, Kinnunen J, Oikarinen K. Factors affecting neurosensory disturbance after mandibular bilateral sagittal split osteotomy. J Oral Maxillofac Surg. 2000 Nov;58(11):1234-9; discussion 1239-40. doi: 10.1053/joms.2000.16621. PMID 11078134
- [Derived] Malkoc Y, Gulsever S, Uckan S. Change in taste sensation after orthognathic surgery. Clin Oral Investig. 2024 Apr 1;28(4):237. doi: 10.1007/s00784-024-05626-1. PMID 38558265
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/26935213/
- Available data/document: Individual Participant Data Set — https://pubmed.ncbi.nlm.nih.gov/26935213/
- Available data/document: Individual Participant Data Set — https://pubmed.ncbi.nlm.nih.gov/11078134/